CLINICAL TRIAL: NCT03329391
Title: A Prospective Study on the Psychosocial Characteristics and Non-pharmacological Intervention of Patients With Treatment-resistant Depression
Brief Title: Psychosocial Characteristics and Non-pharmacological Intervention of Patients With Treatment-resistant Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Shin Kong Wu Ho-Su Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 201612198RINB
Record Dates: First submitted 2017-10-12; First posted 2017-11-06 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2020-06

CONDITIONS: Treatment-resistant Depression
Keywords: Psychosocial model,nursing intervention
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The intervention group will receive a 8-week nurse-led psychosocial care group,which involve 90 minutes session every week.
  Interventions: Behavioral: Nurse-led cognitive-behavioral-based group intervention
- Control Group (No Intervention): The control group will receive usual care, which refers to the pharmacological therapy provided by psychiatrists in the Psychiatric Department.

INTERVENTIONS:
Behavioral: Nurse-led cognitive-behavioral-based group intervention — The intervention focused on the following topics of symptom awareness(i.e. provision of literacy in depression and stress), stress management, lifestyle restructuring and emotional self-care. These topics have been integrated as four major domains for discussions in the eight-weekly sessions. Each session starts with open discussion for participants' daily concerns to activate group dynamics, followed by second part of domain-oriented discussions, and then the third part of session review and homework reminder.
  Arms: Intervention Group

SUMMARY:
Pharmacotherapy and psychotherapy, effective management strategies for treatment-resistant depression are limited and yet to be developed. However, nursing interventions focusing on adherence enhancement, symptom reduction, and stress management may be strategic for a better disease management. This study aimed to define the rarely-studied concept of TRD under the cultural context of Taiwan and to identify new feasible and complementary treatment model from nursing perspectives. The project had established important basis on the descriptions of psychosocial features and need assessment of people with TRD over psychiatrist's validation. The findings also built up a cultural-specific non-pharmacological intervention module for effective TRD management in Taiwan. The nursing model of TRD management will further promote the development of integrative depression care in the future and complement current modalities, while providing important evidence-based information for future research and services.

DETAILED DESCRIPTION:
The three-year pioneering project began with observing the psychosocial characteristics and demographic profile of a group of TRD cohort, followed by validating the cultural meanings and recovery constructs of TRD through professional and lay focus groups in the first year. In the second to third year, we examined the effectiveness of a 8-week, nurse-led psychosocial intervention with group approach in a randomized control trial (RCT) compared to the controls receiving usual care with three follow-ups. Detailed psychiatric assessment and study interviews have been performed at baseline, 3, 6, and 9 months after the intervention by a senior psychiatrist and a research assistant using standardized operation forms.Structured measurements have been utilized to collect primary outcome variables of psychological distress, suicide risk and resilience as well as secondary outcome measures of quality of life, community reintegration level, perceived satisfaction, and main clinical variables (e.g., treatment adherence, service use such as ER/OPD attendance or hospitalization days). The control group receives usual care of pharmacological therapy provided by the psychiatrists in the Psychiatric Department of the study hospital in northern Taiwan.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 20-85 ;
2. To be diagnosed with Major Depressive disorder or Bipolar II disorder;
3. Failed to respond to at least three weeks of two antidepressant trials ;
4. Able to communicate with Mandarin or Taiwanese ;
5. No severe or foreseeing cognitive impairment during study period judged by the co-PI；
6. Willing to sign the informed consent.

Exclusion Criteria:

1. Unable to cooperate due to psychiatric symptom disturbance ;
2. Unwilling to provide most information in the questionnaire ;
3. Severely suicidal during study period

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2018-01-09 (Actual); Primary Completion 2020-09-22 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Change of score of the Brief Symptom Rating Scale(BSRS-5) for psychological distress level | Baseline assessment and follow up sessions on 3,6, and 9 months
  The full scale contains five items of psychopathology: (1) anxiety; (2) depression; (3) hostility; (4) interpersonal sensitivity: inferiority; and (5) insomnia. An extra question "Do you have any suicide ideation?" is added at the end of the scale. It is a 5-item Likert scale (scores of 0 to 4) for assessment of psychological distress level by self-report of by interview. The rating of symptoms is based on a 5-point scale: 0, not at all; 1, a little bit; 2, moderately; 3, quite a bit; 4, extremely. Total score will be calculated based on the 5 questions with a maximum score of 20, where a higher score indicates higher level of psychological distress and poorer mental health status in the past week.
The change of score in 9-item Concise Mental Health Checklist (CMHC-9) for suicide risk assessment | Baseline assessment and follow-up session on the 9th month
  The CMHC-9 is consisted of 9 items assessing psychopathgology (5 items) and suicide risk (4 items). The five item evaluated recent mental distress, lending the measurement from the BSRS-5, i.e., insomnia, anxiety, hostility, depression, and inferiority. The four items reflecting several key suicide risk factors, including lifetime suicide attempt, future suicide intent, alcohol or drug abuse history, and lack of social support. Each item was rated by 0/1, indicating the existence of each symptom, with a total score ranging from 0 to 9. The higher the score, the higher the risk of suicide. The cutoff at 4 points indicates a higher overall suicide risk among clinical or community population.
Change of score in Brief Resilience Coping Scale (BRCS) for tendencies to cope with stress | Baseline assessment and follow up sessions on 3,6, and 9 months
  It is a 4-item measurement tool designed to assess the ability of an individual to cope with stress in a resilient fashion. The response consists of five options at which 1 means the statement "does not describe you at all" and 5 means "it describes you very well". The score is then added up.Among general public, the score of 4-13 indicates low resilient copers; 14-16 indicates medium resilient copers; and 17-20 indicates high resilient copers. However, the scores will undergo validation among a cohort of TRD patients in this study.

SECONDARY OUTCOMES:
Community Integration Questionnaire-Revised (CIQ-R) for the participants' level of community integration | Follow up sessions on 3, 6, and 9 months
  CIQ-R consists of four domains: home integration, social integration, productivity, andelectronic social networking score. The scale contains 18 items. The home integration subscale is made up of 5 items at which each item is scored from 0-2, where 2 indicates highest degree of integration. The Social Integration subscale consists 6 items with the same scoring method mentioned above. The productivity subscale consists of 4 questions with a total points of 7. The electronic social networking subscale consists of 3 questions with a total points of 6. Scores of these subscales are then added up as an overall CIQ score. Maximum score is 35, which represents maximum community reintegration.
EQ-5D questionnaire for quality of life | Follow up sessions on 3, 6, and 9 months
  The EQ-5D is a self-completed questionnaire which contains five dimensions: mobility, self-care, usual activities, pain-discomfort, and anxiety-depression. The level of function in each dimension is classified into three degrees of disability, which is level 1(no disability), level 2(moderate disability), and level 3(severe disability). These responses will then generate a 5-digit descriptor ranging from 1-1-1-1-1 indicating perfect health to 3-3-3-3-3 indicating worth possible state. It is accompanied by a visual analogue scale (EQ-VAS) to assess perceived health conditions, which ranges from 0 (worst imaginable health state) to 100 (best imaginable health state).

CONTACTS AND LOCATIONS:
Overall Officials: Chia-yi Wu, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- Chia-Yi Wu, Taipei, Taiwan

REFERENCES:
- See also: Researcher's profile — https://scholars.lib.ntu.edu.tw/cris/rp/rp06469/information.html